CLINICAL TRIAL: NCT01355029
Title: A Pilot Study of the Evaluation of the Family Informal Caregiver Stroke Self Management (FICSS) Research Project: Impact on Caregiver Psychosocial, Emotional and Health Needs
Brief Title: Evaluation of the Stroke Caregiver Education and Support Program
Acronym: FICSS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: March of Dimes, Canada (Other)
Collaborators: Hamilton Health Sciences Corporation (Other)
Responsible Party: Principal Investigator, Gail Mores, Director, National and Provincial Programs, March of Dimes, Canada
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: OSN1101-000119; 10-668 (Other: Hamilton Health Sciences McMaster University REB)
Record Dates: First submitted 2011-05-13; First posted 2011-05-17 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2016-03

CONDITIONS: Stroke
Keywords: Stroke caregivers; Family Caregivers; Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Stroke Caregiver Education and Support Program — 4 week program offered weekly over a 4 week period. Each session is a 2 hour small group guided discussion on the topic area facilitated by 2 trained facilitators. The topics are: Program Introduction, sharing Caregiving Stories and an introduction to Self Management; Community Connections; Session 3 and 4 are chosen by the participants during session 1 from 6 possible options: Communication in your relationship; Cognition, Memory and Personhood; Dealing with your Emotions; Managing your Stress; Changing roles in your relationships and How to be Caregiver Smart?
  Other Names: FICSS Program

SUMMARY:
The study will be evaluating to a 4 week education and support program for stroke caregivers. The 4 week program will provide education, information, and strategies for dealing with areas that caregivers may find challenging in their caregiving role. The study will evaluate the effectiveness of the program to decrease the caregiver's stress, strain and burden, increase the caregiver's knowledge of strategies and community services and increase their role satisfaction as a stroke caregiver and quality of life two weeks after the program and 6 months after the program.

DETAILED DESCRIPTION:
The modules in the program are: 1) Program Introduction, sharing Caregiving Stories and an introduction to Self Management; 2) Community Connections; Session 3 and 4 are chosen by the participants during session 1 from 6 possible options: Communication in your relationship; Cognition, Memory and Personhood; Dealing with your Emotions; Managing your Stress; Changing roles in your relationships and How to be Caregiver Smart? The programs provides education, information and strategies to deal with the areas that caregivers struggle with as caregivers in order to help them feel better able to prepared to manage as caregivers. Also, the investigators also hope to develop some beginning understanding of when is the best time to provide the program to stroke caregivers to be most helpful to them in their caregiving role.

ELIGIBILITY:
Informal unpaid family stroke caregivers

Inclusion Criteria:

Informal unpaid family stroke caregivers

* 18 years of age or older;
* Have provided care to stroke survivor within the home for at least 2 months;
* Have the ability to communicate in English;
* Live within Central South Ontario Stroke Region or the West GTA Stroke Region.

Exclusion Criteria:

Caregivers who:

* Paid to provide care;
* Are friends who provide care to stroke survivor;
* Are providing palliative care to stroke survivor within the home.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2011-02; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Change in Baseline Bakas Caregiving Outcome Scale at 2 Weeks and 6 Months post Intervention | Baseline, 2 weeks and 6 months Post Intervention
  12 item self report instrument using a 7 point Likert scale 4 designed to measure changes in post stroke caregiver family life changes in the areas of social functioning, subjective well being and physical health,financial well-being, physical functioning, general health, roles in life and level of energy. The revised scale has demonstrated internal consistency reliability of 0.90 and construct validity of 0.66 5. The scale measures both the positive and negative aspects of caregiving with an emphasis on social consequences.

SECONDARY OUTCOMES:
Change in Baseline Oberst Caregiving Burden Scale at 2 Weeks and 6 Months Post Intervention | Baseline, 2 weeks and 6 months post intervention
  15 item self report instrument using a 5 point Likert scale to evaluate caregiver perceptions of the time and difficulty associated with 15 tasks performed in caring for recovering family members. It has been validated in cancer and stroke caregiver populations. It has demonstrated internal consistency reliability of 0.90 - 0.94 and validity of between 0.61 to 0.82 in stroke caregivers.
Open Ended Focus Group Interview to assess impact of program weeks and 6 months post intervention | 2 weeks and 6 months post Intervention
  The questions will be designed to assess the impact on the stroke caregiver; perceived improvement in problem solving abilities; increased awareness and usage of community services; any indirect influence on the stroke survivor; timing of the intervention; and evaluation of the FICSS project.
Caregiver Baseline/Stroke Survivor Baseline Questionnaire | Baseline
  Caregiver Baseline/Stroke Survivor Baseline Questionnaire is a 26 item questionnaire that collects socio-demographic and health related information of the stroke survivor and caregiver. The questionnaire is an adaptation of the one developed by Dr. Jill Cameron to include socio-demographic and health related information on the stroke survivor. The original questionnaire has been utilized in her initial and ongoing research in her "Timing it Right Framework" for stroke caregivers. Permission has been granted by Dr. Cameron to utilize the questionnaire for the study.

CONTACTS AND LOCATIONS:
Overall Officials: Gail Mores, B.Sc. Rec., Principal Investigator — March of Dimes, Canada
Locations (1):
- Hamilton Health Sciences, Hamilton, Ontario, Canada